CLINICAL TRIAL: NCT02141373
Title: Effectivenes of Cyanoacrylate (Glubran 2®) in Reducing Seroma Formation in Breast Cancer Patients Post-Axillary Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Mahmoud Al-Masri, Chairman, Department of Surgery, King Hussein Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRT-CTU-0912/03 Version 5.0
Record Dates: First submitted 2014-04-09; First posted 2014-05-19 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: seroma; axillary; dissection
MeSH Terms: conditions — Breast Neoplasms; Seroma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glubran 2 (Experimental): Glubran 2 will be used at end of surgery
  Interventions: Device: Glubran 2
- Standard Surgery (No Intervention)

INTERVENTIONS:
Device: Glubran 2
  Arms: Glubran 2

SUMMARY:
Glubran 2 as a surgical glue maybe effective in reducing seroma formation post axillary dissection in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* The Patient should be above 18 years old
* The Patients has Node positive breast cancer
* The Patient is eligible for axillary dissection in addition to a surgical intervention for the primary tumor
* Patients whose sentinel lymph nodes test positive during surgery.
* The patient is willing to sign an informed consent to participation

Exclusion Criteria:

* Platelet count is less than 100000
* Obese patients with a BMI of more than 35
* Patients who need immediate breast reconstruction surgery
* Patients who are receiving anticoagulation therapy or have coagulation disorders
* Pregnant or lactating patients
* Patients who are on steroid therapy
* Patients who received chest radiotherapy
* Patients who received neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Total drainage volume | 3 months
Total seroma aspirate volume | 3 months

SECONDARY OUTCOMES:
Adverse events | 3 months
Duration of fluid drainage | 3 months
Time to drain removal | 3 months
Number of seroma aspirations | 3 months
Additional costs incurred due to the need of aspirations | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Al Masri, MD, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

REFERENCES:
- [Derived] Al-Masri M, Alawneh F, Daoud F, Ebous A, Hamdan B, Al-Najjar H, Al-Masri R, Abufara M. Effectiveness of Cyanoacrylate in Reducing Seroma Formation in Breast Cancer Patients Post-Axillary Dissection: A Randomized Controlled Trial. Front Oncol. 2021 Jan 25;10:580861. doi: 10.3389/fonc.2020.580861. eCollection 2020. PMID 33569343